CLINICAL TRIAL: NCT01815125
Title: Ondansetron for Pediatric Mild Traumatic Brain Injury; a Pilot Randomized Controlled Trial.
Brief Title: Ondansetron for Pediatric Mild Traumatic Brain Injury
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZOF2013; 9427-c2686-28c (Other: Health Canada)
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2014-02

CONDITIONS: Traumatic Brain Injury; Brain Concussion
Keywords: Mild traumatic brain injury; Brain concussion; Post-concussion syndrome; Emergency department; Ondansetron
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Post-Concussion Syndrome; Emergencies | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Experimental): The intervention of interest will be the administration of one dose of oral ondansetron in the emergency department. The dosage will be 8 mg.
  Interventions: Drug: Ondansetron
- Placebo (Placebo Comparator): The control group will receive a similar looking/ tasting pill of placebo.
  Interventions: Drug: PLacebo

INTERVENTIONS:
Drug: Ondansetron — The intervention of interest will be the administration of one dose of oral ondansetron in the emergency department. The dosage will be 8 mg.
  Other Names: Zofran
  Arms: Ondansetron
Drug: PLacebo — placebo
  Arms: Placebo

SUMMARY:
Background: Most patients suffering from mild Traumatic Brain Injury (mTBI) present persistent symptoms at one week post injury. A systematic review showed a paucity of studies for short term outcomes following mTBI. Among potential treatments for mTBI, ondansetron has shown promising results based on clinical experience and a single retrospective study. Objectives: The primary objective of this pilot study is to determine the feasibility of a randomized controlled trial evaluating the effect of ondansetron to decrease post concussion symptoms at one week following mTBI in children. More specifically, this pilot study will evaluate the proportion of participants who complete assessment at one week following intervention. Method: This will be a randomized, double blinded, controlled trial performed among children aged between 8 and 17 years old who sustained a mTBI in the previous 24 hours. Participants visiting the emergency department will be randomized to receive one dose of either ondansetron or placebo. The primary outcome of interest is defined as an increase from pre-concussion baseline of at least 3 symptoms from the Post Concussion Symptom Inventory (PCSI) one week following trauma. Secondary outcomes will include time to full recovery, mean PCSI score, and outcomes at one month following head trauma. The primary analysis will compare the proportion of participants with persistence of symptoms at one week in both groups. The full study sample size was calculated to have 90% power to detect a decrease in the proportion of persistence of symptoms from 50% to 30% with an alpha value of 0.05. Approximately 126 patients will therefore be recruited in each arm. The investigators plan to recruit 30 participants (10% of the final population) for the pilot study. Expected results: This pilot study should confirm the feasibility of the randomized controlled trial by showing that 90% of the recruited participants provide data on the primary outcome at one week following intervention. On the long term, the investigator expect that ondansetron will decrease the proportion of patients sustaining persistent symptoms of concussion from 50% to lower than 30%.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged between 8 and 17 years old. This will be limited to this small spectrum of age to insure better homogeneity in the evaluation of the participants and streamlining of outcome measures. Also, this is the age group for which our measurement tool has been validated.
2. Occurrence of a mTBI as defined by the presence of a head trauma, a Glasgow coma scale of 13 to 15 and at least one of the three following criteria4 :

   * Any period of loss of consciousness.
   * Any loss of memory for events immediately before or after the accident.
   * Any alteration in mental state at the time of the accident (eg, feeling dazed, disoriented).

   And the absence of the following criteria:
   * Post-traumatic amnesia greater than 24 hours.
   * Glasgow Coma Scale < 13, 30 minutes post accident.
3. The trauma occurred in the preceding 24 hours.

Exclusion Criteria:

* 1. Inability to obtain a proper written informed consent (language barrier, absence of a parental authority, developmental delay, intoxication, patient too confuse to consent according to the treating physician).

  2. Known allergic reaction or intolerance to ondansetron. 3. Known rhythm or cardiac problem, or history of sudden death in the proximal family 4. Patients who are taking a medication which could increase the QT interval. 5. Patients who received ondansetron in the previous 24 hours 6. Any abnormality on radiological studies, including any bleeding in the brain or skull fracture.

  7. Multi-system injuries with treatment requiring admission to hospital or procedural sedation in the ED.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Persistence of post concussive symptoms | 1 week post intervention
  Persistence of post concussive symptoms will be defined by an increase from pre-concussion baseline of at least 3 symptoms of the Post Concussion Symptom Inventory (PCSI). The PCSI is a self-report tool evaluating the presence of 25 symptoms (on a 3-point likert scale) for children 8-12 and 26 symptoms on a (7-point likert scale) for children 13-17 years. An increase of two points or more from pre-injury in any symptom is considered clinically significant.

SECONDARY OUTCOMES:
Mean number of PCSI symptoms | one week and month following intervention
Mean number of school days missed | one month following intervention
Number of days of sport activity restriction | 1 month following intervention
Time before full recovery | One month following intervention
  According to the parents
Healthcare utilization | One month following intervention
  Proportion of participants who consulted a health resource.
Side effects | one week and month following intervention
  Side effects will include, in addition to symptoms related to mTBI,proportion of participants who complained of diarrhea or constipation (binary answer).

OTHER OUTCOMES:
Proportion of participants who complete the assessment at one week following intervention | One week following intervention
  the main objective of the pilot study is to evaluate the feasibility of the randomized controlled trial. Accordingly, the primary outcome of the pilot study will be the proportion of participants who complete the assessment at one week following intervention
Proportion of eligible children who were not included | At baseline
  This is the proportion of eligible children who were not included and reasons for non-inclusion.
Compliance with study medication | One week following intervention
  Proportion of patients who tolerated their medication and proportion of patients randomized to the control group who received ondansetron

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Gravel, MD, Principal Investigator — CHU Sainte-JUstine, University of Montreal
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada